Informed Consent Document Attention, Teleconferencing and Social Anxiety

Date: 12/02/2020

Identifiers: NCT04729803 Unique Protocol ID: STUDY00000106

Title of the Project: Investigating Attentional Processes: Teleconferencing and Social Anxiety Part 1

Principal Investigator: Mikael Rubin, Graduate Student, UT Austin

Faculty Advisor: Michael J. Telch, Ph.D., Professor of Psychology & Psychiatry, UT Austin

# **Consent to Participate in Research**

## Invitation to be Part of a Research Study

You are invited to be part of a research study. This consent form will help you choose whether or not to participate in the study. Feel free to email us if anything is not clear in this consent form.

## What is the study about and why are we doing it?

The purpose of this study is to understand how people pay attention during zoom calls.

Teleconferencing can elicit some social anxiety and influence who you pay attention to during a call and during an interaction.

#### What will happen if you take part in this study?

If you agree to take part in this study, you will first be asked to complete some questionnaires about your background and how you've been feeling lately.

Depending on your answers to the questionnaires you may then be randomly assigned (like the flip of a coin) to one of the following groups: (a) positive interactions; (b) negative interactions. And be linked to a teleconferencing call where you will be asked to respond briefly to one question that one of the other people asks. You will be asked to do this twice. We are interested in where you are looking during these calls and you will be asked to complete some brief procedures so that we can measure where you are looking. Audio and video will be recorded during these calls.

Based on your responses you will have the option to enroll in a second part of this study where you would do more teleconferencing interactions to help reduce social anxiety symptoms.

## How long will you be in this study and how many people will be in the study?

Participation in this study will last approximately 30 minutes. We expect to enroll 2,000 participants for this study.

# What risks and discomforts might you experience from being in this study?

The risks are no greater than those experienced in daily life.

#### How could you benefit from this study?

There are no direct benefits to participating. There are potential benefits to society resulting from your participation in this study. These include providing new knowledge on attention social anxiety and teleconferencing.

#### What will happen to the data we collect from you?

As part of this study we will collect basic personal information such as your sex, age, ethnicity/race, current living arrangements and contact information. We will also obtain important data from well-established questionnaire measures rating your social anxiety. We will collect audio and eye movement data related to your interactions during the teleconferencing calls.

# How will we protect your information?

We will protect your information by making sure that your name or any other information that can directly identify you are stored in a secure HIPPA compliant platform separately from data collected from you as part of the study. Information about you may be given to the following organizations: Representatives of UT Austin and the UT Austin Institutional Review Board. We may share your data with other researchers for future research studies that may be similar to this study or may be very different. The data shared with other researchers will not include information that can directly identify you. Last, we plan to publish the results of this study. To protect your privacy, we will not include any information that could directly identify you.

## What will happen to the information we collect about you after the study is over?

We will keep your data to use for future research. All identifiable data (including the audio data) will be destroyed once analyses have been completed.

Please check this box if you consent to have your name and email retained after completion of the study for the purpose of being contacted for future research studies.

[check box]

# How will we compensate you for being part of the study?

If you are in the undergraduate research pool you will receive up to 1 credit for participation in this part of the study.

If you are not participating for course credit you will be entered into a drawing for \$10 after you complete this part that will be sent digitally through Venmo or Paypal. There will be five drawings for \$10.

# What other choices do you have if you do not take part in this study?

Should you choose not to participate in this study if you are in the undergraduate research pool then you can complete the alternative writing assignment. If you are not in the undergraduate research pool you can simply exit out of the survey at any time.

# Your Participation in this Study is Voluntary

It is totally up to you to decide to be in this research study. Participating in this study is voluntary. Your decision to participate will not affect your relationship with The University of Texas at Austin. You will not lose any benefits or rights you already had if you decide not to participate. Even if you decide to be part of the study now, you may change your mind and stop at any time. You do not have to answer any questions you do not want to answer. If you decide to withdraw before this study is completed, data that could reveal your identity (i.e., name, email, etc.) will be destroyed but non-identifiable data will be retained indefinitely.

#### **Contact Information for the Study Team**

If you have any questions about this research, you may contact:

Mikael Rubin, Phone: 646-685-4681; Email: mikaelrubin@utexas.edu

Dr. Michael J. Telch; Phone: (512) 967-1094; Email: DrTelch@gmail.com

# Contact Information for Questions about Your Rights as a Research Participant

If you have questions about your rights as a research participant, or wish to obtain information, ask questions, or discuss any concerns about this study with someone other than the researcher(s), please contact the following:

The University of Texas at Austin Institutional Review Board

Phone: 512-232-1543

Email: irb@austin.utexas.edu

Please reference study number 106.

# **Session Recordings**

Video and Audio of your teleconferencing interactions will be recorded. They will be stored separately from any other study information using secure data storage services. Please acknowledge that you understand and accept that the interactions will be recorded.

[check here]

#### **Your Consent**

By clicking "I consent" below, you are agreeing to be in this study. If you do not agree to be in this study, simply close your browser window.

I understand what the study is about and my questions so far have been answered. I agree to take part in this study by checking the box below.

[click here]

Title of the Project: Investigating Attentional Processes: Teleconferencing and Social Anxiety Part 2

Principal Investigator: Mikael Rubin, Graduate Student, UT Austin

Faculty Advisor: Michael J. Telch, Ph.D., Professor of Psychology & Psychiatry, UT Austin

# **Consent to Participate in Research**

## Invitation to be Part of a Research Study

You are invited to be part of a research study. This consent form will help you choose whether or not to participate in the study. Feel free to email us if anything is not clear in this consent form.

## What is the study about and why are we doing it?

The purpose of this study is to understand whether practicing interactions during teleconferencing can help reduce social anxiety.

#### What will happen if you take part in this study?

If you agree to take part in this study, you will be randomly assigned (like the flip of a coin) to one of the following three intervention groups: (a) attention guidance + exposure; (b) attention control + exposure; or (c) exposure alone. You may be asked to wait for 1-week before starting.

- 1. Information component (15 minutes). Prior to beginning the intervention you will see a pre-recorded researcher discuss social anxiety, the intervention, what you will be asked to do
- 2. Intervention sessions (45 minutes each). You will have the chance to complete up to 4 intervention sessions within a two-week period from the first time you receive the link. Each time you complete one intervention session you will be sent a new link to complete another session.
- 3. Follow-Up Assessments (15 minutes each). In order to determine the extent to which the intervention was helpful, immediately following your last intervention session two weeks after completing the intervention you will be asked to complete a separate online follow-up. During the follow-ups, you will be asked to complete the same assessments as part 1 of the study.

We are interested in where you are looking during these teleconferencing calls and you will be asked to complete some brief procedures so that we can measure where you are looking. Audio and video will be recorded during these calls.

# How long will you be in this study and how many people will be in the study?

Participation in this study will last up to 4 weeks. Your participation will require from 1 hour up to 4 hours total. We expect to enroll 100 participants for this part of the study.

## What risks and discomforts might you experience from being in this study?

The risks are no greater than those experienced in daily life.

## How could you benefit from this study?

There are no direct benefits from the study. There are potential benefits to society resulting from your participation in this study. These include providing new knowledge on attention social anxiety and teleconferencing.

# What will happen to the data we collect from you?

As part of this study we will collect basic personal information such as your sex, age, ethnicity/race, current living arrangements and contact information. We will also obtain important data from well-established questionnaire measures rating your social anxiety. We will collect audio and eye movement data related to your interactions during the teleconferencing calls.

#### How will we protect your information?

We will protect your information by making sure that your name or any other information that can directly identify you are stored in a secure HIPPA compliant platform separately from data collected from you as part of the study. Information about you may be given to the following organizations: Representatives of UT Austin and the UT Austin Institutional Review Board. We may share your data with other researchers for future research studies that may be similar to this study or may be very different. The data shared with other researchers will not include information that can directly identify you. Last, we plan to publish the results of this study. To protect your privacy, we will not include any information that could directly identify you.

#### What will happen to the information we collect about you after the study is over?

We will keep your data to use for future research. All identifiable data (including the audio data) will be destroyed once analyses have been completed.

# How will we compensate you for being part of the study?

If you are completing this study for SONA research credit you will receive credit based on the amount of time you spend completing the study. Each component of the study takes a different amount of time. Based on the amount of time you spend (i.e. components you complete) you will receive the equivalent credits. If you spend 1 hour participating, you will receive 1 credit, and so on.

If you are not participating for course credit you will be entered into a drawing for \$50 after you complete this part that will be sent digitally through Venmo or Paypal. There will be five drawings for \$50.

## What other choices do you have if you do not take part in this study?

Should you choose not to participate in this study but would like information about alternative treatment options, you can find referral resources at the end of the study – or you can reach out to study staff who will provide you with a list of treatment referral resources.

#### **Your Participation in this Study is Voluntary**

It is totally up to you to decide to be in this research study. Participating in this study is voluntary. Your decision to participate will not affect your relationship with The University of Texas at Austin. You will not lose any benefits or rights you already had if you decide not to participate. Even if you decide to be part of the study now, you may change your mind and stop at any time. You do not have to answer any questions you do not want to answer. If you decide to withdraw before this study is completed, data that could reveal your identity (i.e., name, phone number, email, etc.) will be destroyed but non-identifiable data will be retained indefinitely.

## **Contact Information for the Study Team**

If you have any questions about this research, you may contact:

Mikael Rubin, Phone: 646-685-4681; Email: mikaelrubin@utexas.edu

Dr. Michael J. Telch; Phone: (512) 967-1094; Email: <a href="mailto:DrTelch@gmail.com">Dr. Michael J. Telch@gmail.com</a>

#### Contact Information for Questions about Your Rights as a Research Participant

If you have questions about your rights as a research participant, or wish to obtain information, ask questions, or discuss any concerns about this study with someone other than the researcher(s), please contact the following:

The University of Texas at Austin Institutional Review Board

Phone: 512-232-1543

Email: irb@austin.utexas.edu

Please reference study number 106.

#### **Session Recordings**

Your teleconferencing interactions will be recorded. They will be stored separately from any other study information using secure data storage services. Please acknowledge that you understand and accept that the interactions will be recorded.

[check here]

#### **Your Consent**

By signing below, you are agreeing to be in this study. You can download a copy of this document for your records. We will keep a copy with the study records. If you have any questions about the study after you sign this document, you can contact the study team using the information provided above. If you do not agree to be in this study, simply close your browser window.

| I understand what the | study is about a | nd my questioi | ns so far have | e been answere | d. I agree to |
|---|---|---|---|---|---|
| take part in this study. | | | | | |

| Typed Subject Name | |
|----------------------|------|
| Electronic Signature | Date |